CLINICAL TRIAL: NCT04007211
Title: A Randomized, Multi-center, Evaluator and Subject Blind, Active-controlled, Parallel, Medical Device Pivotal Clinical Study to Assess the Anti-adhesive Effect and Safety of ABT13107 Compared to Hyalobarrier Applied to Postoperative Intrauterine
Brief Title: Pivotal Clinical Study to Assess the Anti-adhesive Effect and Safety of ABT13107 Applied to Postoperative Intrauterine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT10-KR16IUA705
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Adhesion of Uterus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABT13107 (Experimental)
  Interventions: Device: ABT13107
- Hyalobarrier (Active Comparator)
  Interventions: Device: Hyalobarrier

INTERVENTIONS:
Device: ABT13107 — Dose: 3mL, maximum 10mL
  Arms: ABT13107
Device: Hyalobarrier — Dose: 10mL
  Arms: Hyalobarrier

SUMMARY:
This study is intended to evaluate the efficacy and safety of ABT13107 compared to Hyalobarrier applied to postoperative intrauterine.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged from 19 to 70
* Those who are scheduled for hysteroscopy to treat the following diseases: submucosal myomas, endometrial polyps, intrauterine adhesion etc.

Exclusion Criteria:

* Those who will apply other intrauterine device rather than investigational device during the study period.

Ages: 19 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Incidence of intrauterine adhesion | 4 weeks
  Incidence rate of intrauterine adhesion after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee DY, Lee SR, Kim SK, Joo JK, Lee WS, Shin JH, Cho S, Park JC, Kim SH. A New Thermo-Responsive Hyaluronic Acid Sol-Gel to Prevent Intrauterine Adhesions after Hysteroscopic Surgery: A Randomized, Non-Inferiority Trial. Yonsei Med J. 2020 Oct;61(10):868-874. doi: 10.3349/ymj.2020.61.10.868. PMID 32975061